CLINICAL TRIAL: NCT02938884
Title: Investigation of Non-Invasive Hydration Monitoring With Smart Water Bottle to Increase Fluid Intake in Patients With Nephrolithiasis and Low Urine Volume
Brief Title: Hidrate Me Smart Water Bottle Use in Patient With Nephrolithiasis
Acronym: HidrateMe
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: URO-2016-25230
Record Dates: First submitted 2016-10-12; First posted 2016-10-19 (Estimated); Last update posted 2021-07-14 (Actual); Status verified 2021-07

CONDITIONS: Nephrolithiasis; Low Urine Volume
MeSH Terms: conditions — Nephrolithiasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HidrateSpark Water Bottle (Active Comparator): Patients meeting the eligibility criteria who are interested in participating in the study and randomized to receive the "HidrateSpark" water bottle be given one at no cost. They will download the associated free software application to their smartphone and be given education in the outpatient setting regarding how to use the system.
  All subjects in both cohorts will be provided the same questionnaire on two occasions, at the beginning and end of the trial, to determine their attitudes about fluids and potentially identify barriers to maintaining adequate hydration status (Appendix A). Additionally, standard information from the medical record including demographics, occupation, medical history and medications will be recorded.
  Interventions: Device: HidrateSpark Water Bottle
- No Smart water bottle (No Intervention): All subjects in both cohorts will be provided the same questionnaire on two occasions, at the beginning and end of the trial, to determine their attitudes about fluids and potentially identify barriers to maintaining adequate hydration status (Appendix A). Additionally, standard information from the medical record including demographics, occupation, medical history and medications will be recorded.

INTERVENTIONS:
Device: HidrateSpark Water Bottle — HidrateSpark water bottle is a smart water bottle that glow when its time to drink water. It is run through an app on a smart phone
  Arms: HidrateSpark Water Bottle

SUMMARY:
The primary objective of this study would be to determine whether utilization of this technology improves adherence to recommended increases in hydration for stone forming patients with low urine volume relative to standard techniques such as education and reading materials. We hypothesize that the addition and utilization of the smart water bottle to standard recommendations will lead to measurable increases 24 hour urine output for affected patients.

DETAILED DESCRIPTION:
Nephrolithiasis is one of the most common and costly diseases in medicine affecting nearly 10% of the population. It is also the most costly urologic disease with an estimated ten billion dollars per year in associated healthcare expenditures towards treating this condition. One of the biggest obstacles in controlling the growing incidence of the disease is better preventative care, especially considering that one third to one half of the patients who have a single stone event will have another stone within the next ten to fifteen years. Despite decades of research on preventative strategies to reduce stone recurrences there are only a handful of dietary and medical treatments with strong evidence supporting their use.

One of the cornerstones of kidney stone prevention is ensuring adequate fluid intake. Without adequate hydration, urinary volume is low which in turn increases super-saturation of all stone forming salts and increases the likelihood of stone formation. The best evidence supporting adequate fluid as a prevention strategy for stones comes from Borghi et al. who performed a 5 year randomized control study and found a 12% recurrence rate in the cohort of patients encouraged to achieve a goal of 2 liters (L) of urine per day compared to a 27% recurrence in the group who was not encouraged to increase fluid intake. Furthermore, the most recent guidelines by both the American Urological Association (AUA) and American College of Physicians (ACP) on medical management of kidney stones advocate a goal urine volume of 2.5 L for all stone formers.

Despite recommendations and evidence supporting its utility as an effective prevention mechanism for stone formers, achieving significant increases in hydration and subsequently urinary volumes remains a considerable clinical challenge. To date, adherence to increased fluid recommendations has been understudied with little data assessing patient compliance specifically for fluid. However, noncompliance with metabolic treatment of nephrolithiasis is common with estimates that only 50% of patients follow recommendations.These rates are similar to rates of noncompliance with recommended care in other chronic medical conditions as well including diabetes, chronic kidney disease, congestive heart failure, and metabolic syndrome.

Recently, mobile health technology has received much attention as a potential aide in helping improve compliance with medically indicated lifestyle and dietary treatments. Early studies using "smart technology" and mobile health applications have shown that implementation of such strategies can not only be beneficial in improving compliance, but also have the potential to lead to sustainable behavioral change. To date, there are no studies looking at mobile health technology as it applies to increasing fluid intake, particularly among stone formers.

Recently, a novel "smart" water bottle called "HidrateSpark" (www.hidratespark.com) developed by researchers at the University of Minnesota has been developed for use as a noninvasive fluid intake monitoring system. The device uses capacitive touch sensing via a sensor extending from the lid to the base, which calculates volume measurements by detecting changes in water levels. Data from the bottle is sent wirelessly to users' smartphones through an application.

This device has significant potential for use particularly among stone former that have demonstrated difficulty increasing their hydration as a part of preventative care. The device would not only allow users the ability to closely monitor their fluid intake throughout the day, it would also engage the patient with reminders to drink periodically throughout the day and stay hydrated. Additionally, fluid intake measurements stored through the associated application have the potential to be used as a novel metric capable of being brought to the provider's attention in order to better assess and guide patient hydration status and identify barriers to achieving hydration goals.

The primary objective of this study would be to determine whether utilization of this technology improves adherence to recommended increases in hydration for stone forming patients with low urine volume relative to standard techniques such as education and reading materials. We hypothesize that the addition and utilization of the smart water bottle to standard recommendations will lead to measurable increases 24 hour urine output for affected patients.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* History of known kidney stone event (radiographic, passed, or treated)
* Documented history of low urinary volume on at least one 24 hour urine analysis (<1.5L) within past 6 months of potential enrollment
* No planned changes to medication based on most recent 24 hour urine analysis

Exclusion Criteria:

* Cognitive impairment
* Lack of smartphone
* Coexisting medical condition that precludes high fluid intake such as chronic kidney disease, congestive heart failure, SIADH.
* Significant voiding dysfunction (i.e. BPH, LUTS, interstitial cystitis, neurogenic bladder, incontinence)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2016-12-05 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline in hydration adherence at 12 weeks, as determined by measurable increase in urine volume | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Michael Borofsky, MD, Principal Investigator — University of Minnesota
Locations (4):
- United States (4):
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - University of Chicago, Chicago, Illinois
  - Indiana University, Bloomington, Indiana
  - Mayo Clinic Rochester, Rochester, Minnesota

REFERENCES:
- Available data/document: Study Protocol — https://oncore.umn.edu/login/